CLINICAL TRIAL: NCT05291611
Title: Smart Sensory Technology in Telepsychotherapy for the Treatment of Obsessive-compulsive Disorder in Children and Adolescents
Brief Title: Smart Sensory Technology in Psychotherapy for Pediatric OCD
Acronym: SSTeP-KiZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Universität Tübingen (Other); University of Hohenheim (Other)
Responsible Party: Principal Investigator, Prof. Dr. Tobias Renner, Prof. Dr. Tobias Renner, Head of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 877/2020BO1
Record Dates: First submitted 2021-12-10; First posted 2022-03-22 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-compulsive Disorder; Children and Adolescents; Cognitive-behavioral therapy; Digital sensory device
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: All participants will be treated with cognitive behavioural therapy during our feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with cbt (Experimental): Treatment for 26 patients with obsessive-compulsive disorder, 14 sessions, each about 90 minutes.
  Interventions: Behavioral: Online-based Cognitive-behavioral Therapy for OCD

INTERVENTIONS:
Behavioral: Online-based Cognitive-behavioral Therapy for OCD — 26 patients with obsessive-compulsive disorder (OCD) receive treatment with cognitive-behavioral therapy. 14 sessions will take place via the internet.
  Other Names: Online-based Psychotherapy

SUMMARY:
Telemedicine interventions enable the improvement of behavioral state-of-the-art treatment of OCD, as therapy can be delivered in the patients' immediate home environment, allowing for more valid symptom actualization. In addition, access to experts is made possible even in rural areas, and the inhibition to seek therapy can be reduced. In a preliminary study, our research group was able to demonstrate the efficiency of using telemedical access. SSTeP-KiZ aims at the further development of telemedical treatment of children with OCD by using sensor technology in the home setting, where most symptoms occur. In this context, relevant emotional states of the patients such as anxiety and stress reactions shall be quantified reliably during the therapy session with exposures by combining different sensor modalities. As a result, the therapy procedure can be immediately and individually adapted to the patient and the situation, thus optimizing the success of the treatment.

Methods: It is planned to establish the therapy system on a sample of 10 healthy children and 5-10 patients with OCD treated at University Hospital of Tübingen. Afterwards we will recruit 26 children with obsessive-compulsive disorder aged 12-18 years to conduct therapy with them. There are 14 weekly therapy sessions via teleconferencing with the children and parents. During the sessions and exposures, patients' field of view is recorded via eye trackers, measures of stress responses via heart rate and pupillometry, and movement measures for approach-avoidance behaviors. Using an AI approach, these indicators are integrated and reported back to the therapist online to optimize the therapy process. Accompanying app-based daily symptoms will also be collected by the children and parents and processed for use in the therapy process. We expect a good feasibility and significant symptom reduction by this therapeutic approach and the chance to make this system usable for broad clinical application.

DETAILED DESCRIPTION:
The main goal of SSTeP-KiZ is the implementation of sensors in the existing telepsychotherapeutic treatment of children and adolescents with obsessive-compulsive disorder. SSTeP-KiZ aims to significantly improve the telepsychotherapeutic treatment options for this group of patients through the use of sensors that can be worn during symptom triggering situations at home in patients' everyday lives, and an analysis and incorporation of the multimodal sensor data into the therapeutic process.

In the medium term, SSTeP-KiZ should enable the use of real-time data on anxiety and stress levels (pupillometry, heart rate, eye tracking) obtained during therapy sessions by the therapist while the patient is still in the therapy session. Thus, even under the conditions of telepsychotherapy, despite the physical absence of the therapist, the individual intensity of the therapy sessions can be directly adjusted. In addition, the compliance and satisfaction of the patients during the accompanied therapy tasks can be directly promoted. Furthermore, the data obtained within the framework of SSTeP-KiZ should also be suitably prepared concerning the children and adolescents and their relatives and, in the sense of therapeutic feedback, suitably visualized to form an additional component of the therapy.

Goals:

A. Development of a prototype for a multisensory therapy system in healthy children and adaptation to mentally ill children with an obsessive-compulsive disorder.

B. Evaluation of the prototype in the context of an internet-based psychotherapy for mentally ill children with an obsessive-compulsive disorder C: Preparations for the introduction of the multisensory therapy system into broad clinical application in the health care system

Sample I: 10 healthy children:

Sample II: 5-10 patients of University Hospital Tübingen with OCD.

Sample III&IV: 6 & 20 children with OCD.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents with obsessive-compulsive disorders
* aged 12 to 18 years
* a primary DSM-5 obsessive-compulsive disorder
* at least one primary caretaker
* German-speaking (child & caretakers)
* family home equipped with broadband internet connection
* written informed consent of the child and its caretakers
* psychiatric comorbidities will be allowed as long as the comorbid disorder does not have a higher treatment priority than OCD (i.e., psychosis, eating disorder and severe depression)
* Medication is allowed if treatment was stable for 6 weeks before diagnostics and will then be taken during the trial.

Exclusion Criteria:

* IQ below 70
* patients do not speak or understand German
* patients have a psychiatric comorbidity or suicidality that makes participation clinically inappropriate
* too seriously ill so that they should be treated in the hospital
* stable social environment, able to support the children adequately during therapy. - drug addiction
* if the family seems to be severely psychologically burdened so that participation in the sessions and support of the children during the trial will not be possible
* no other psychological treatment is allowed
* If reporting side effects or circumstances that make iCBT treatment clinically inappropriate, or if wished by the patients, the patients are excluded from the study and transferred to another more appropriate therapy option.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) - assessment of the change in the handling of the technical equipment during treatment | After week 1, week 7 and week 14
  Patients are to answer a total of 60 questions with 10 questions for each technical device from the system usability scale (SUS), regarding the handling of the technical equipment and to capture the change in it.
Therapy Process Questionnaire (TPQ) - assessing the stability of the therapeutic relationship and possible changes in the treatment process | Weekly after each therapy session, for 14 weeks of therapy
  Patients are to rate how they perceive the therapeutic process.
Client Satisfaction Questionnaire-8 (CSQ-8) | After the last session in week 14 (post treatment)
  We assess participant's perceptions of the value of the treatment they received
Questionnaire for the evaluation of the treatment (FBB) | After the last session in week 14 (post treatment)
  It records how satisfied the participants were with the treatment. We reduced the total number of questions from 20 to 17, as 3 items covered circumstances that did not occur in the context of internet-based therapy.
Change in Health Care Utilization, measured by HCU-Q (Health Care Utilization-Questionnaire) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  Questionnaire to capture costs and time spent on online-based treatments; Health Care Utilization-Questionnaire, change is assessed between baseline and the last session.
Change in Quality of Life: EQ-5D-3L (European Quality of Life Five Dimensions Questionnaire) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  Questionnaire to capture costs and time spent on online-based treatments: Questionnaire to capture costs and time spent on online-based treatments, measured by European Quality of Life Five Dimensions Questionnaire Three Level Version (EQ-5D-3L).
Change in costs spent on online interventions: CIIQ (Caregiver Indirect and Informal Care Cost Assessment Questionnaire) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  Questionnaire to capture costs and time spent on online-based treatments: Caregiver Indirect and Informal Care Cost Assessment Questionnaire (CIIQ)
Change in affinity for technology (TA-EG) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  Technology Affinity Questionnaire (TA-EG): The TA-EG can be answered by patients and their parents and contains 19 items. It measures the attitude towards and use of electronic devices.
Change in attitudes toward and satisfaction with telemedicine psychotherapy (EZtP) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  Questionnaire on the Attitude and Satisfaction of Telemedicine Psychotherapy (EZtP). The EZtP is a self-developed questionnaire that measures attitudes to and satisfaction with telemedicine psychotherapy. It can be answered by both the adolescents and the parents.
Barriers to Treatment Participation Scale (BTPS) | Once after treatment (t1, after 14 weeks)
  The Barriers to Treatment Participation Scale, is a 44 item rating of how much parents agree with statements about their expectancies of barriers to treatment participation for their child, using a 5-point Likert scale (1=totally disagree, 5= totally agree).
Measures of feasibility: Manual Rating Form (MRF) | Once after treatment (t1, after 14 weeks)
  The Manual Rating Form (MRF) is used to assess feasibility of the manual.
Measures of feasibility: Summary Therapist Feedback Form (STFF) | Once after treatment (t1, after 14 weeks)
  The Summary Therapist Feedback Form (STFF) is used to assess the ease of manual implementation completed after each case.
Implementation and satisfaction questionnaire for the children | Once after treatment (t1, after 14 weeks)
  We designed an implementation and satisfaction questionnaire for the children. It covers the subject's dosage, quality, adaption, responsiveness and program differentiation.
Implementation and satisfaction questionnaire for the parents | Once after treatment (t1, after 14 weeks)
  We designed an implementation and satisfaction questionnaire for the parents. It covers the subject's dosage, quality, adaption, responsiveness and program differentiation.
Implementation and satisfaction questionnaire for the therapist | Once after treatment (t1, after 14 weeks)
  We designed an implementation and satisfaction questionnaire for the therapist. Questions regarding whether the intervention was being delivered as written (adherence) and the representativeness of the participants (reach) were implemented in the therapist's questionnaire covering questions like "The psychoeducation/relapse prophylaxis/exposure sessions were carried out as planned." and a checklist regarding information e.g. about the socioeconomic status, age, gender or IQ.

SECONDARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The CY-BOCS is a clinician-administered instrument that evaluates obsessions and compulsions separately on time consumed, distress, interference, resistance, and control. A score higher than 16 describes clinical relevant obsessive-compulsive symptoms. The short form of the CY-BOCS is conducted daily on the app as part of the mobile assessment.
Children's Global Assessment Scale (CGAS) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The CGAS is a clinician's rating of the patient's overall level of functional strain.
Clinical Global Impressions-Improvement (CGI-I) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The CGI-I is used to assess overall clinical improvement based on symptoms observed and impairment reported. The clinical-rated scale has been used successfully in patients with OCD.
Clinical Global Impressions-Severity (CGI-S) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  Is a clinical rating of symptom severity. The CGI-S correlates strongly with the CY-BOCS total score in pediatric OCD patients, and is widely used and has been shown to be treatment sensitive.
Children's DIPS Open Access: Diagnostic Interview in Childhood and Adolescent Mental Disorders (Kinder-DIPS) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The Kinder-DIPS is a structured clinical interview for the diagnosis of mental disorders. There is a child version and a parent version. Both, the child version and the parent version, are performed.
Brief Self-Control Scale | After week 1, week 7 and week 14
  Patients will be given questions concerning self-control (Brief Self-Control Scale, German Version (Sproesser et al., 2011))
Self-efficacy | After week 1, week 7 and week 14
  Patients answer questions regarding self-efficacy according to the questionnaire of Schwarzer & Jerusalem (1999).
Coping strategies | After week 1, week 7 and week 14
  Patients answer questions regarding coping strategies according to the questionnaire of Schwarzer & Jerusalem (1999).
Self-regulation | After week 1, week 7 and week 14
  Patients answer questions regarding self-regulation according to the questionnaire of Schwarzer & Jerusalem (1999).
Procrastination | After week 1, week 7 and week 14
  Patients answer questions regarding procrastination according to the questionnaire of Schwarzer & Jerusalem (1999).
Child Behavior Checklist (CBCL) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The Child Behaviour Checklist (CBCL/6-18R) is used to record behavioural problems, emotional problems, somatic complaints as well as social competences of children and adolescents of school age from the parents' point of view.
Youth Self-Report (YSR) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The YSR/11-18R (youth version) was derived directly from the CBCL and allows an assessment of the largely identical characteristics from the perspective of adolescents.
Child Obsessive-Compulsive Impact Scale (COIS-RC) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The COIS-RC Culture includes a parent and a child report. It is a 33-item questionnaire designed to assess the impact of OCD symptoms on the psychosocial functioning of children and adolescent in home, social, and academic environments.
Fair Intelligence Test (CFT 20-R) | Baseline (t0) before treatment
  The CFT 20-R records the basic intelligence according to the general fluid ability.
Questionnaire for self-assessment of depressive disorders (DISYPS-III SBB- DES) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The SBB-DES (DYSIPS-III) is a self-report questionnaire for adolescents (11 to 18 years) and part of the Diagnostic System for Mental Disorders according to ICD-10 and DSM-5 for children and adolescents. It records the different symptoms of a depressive disorder, the extent of distress and the competencies of the adolescent.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The SCARED is a psychometrically sound child- and parent-report questionnaire which assesses the presence of DSM-IV anxiety symptoms.
Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents (KIDSCREEN) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The questionnaires can be used to assess the subjective health and well-being of children and adolescents aged 8 to 18 years. A corresponding parent version is available for parents.
Ulm Quality of Life Inventory for Parents of Chronically Ill Children (ULQUIE) | Baseline (before treatment (t0)) and after treatment (t1, after 14 weeks)
  The ULQUIE was used to record the quality of life of the parents.
Affect questionnaire | Daily after each therapy session (approximately 5-10 minutes), for a time period of 14 weeks of therapy
  The emotional state of the patients is recorded daily by the app (ambulatory assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Conzelmann, Prof., Principal Investigator — University Hospital Tübingen; Tobias J Renner, Prof., Principal Investigator — University Hospital Tübingen
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollmann K, Allgaier K, Hohnecker CS, Lautenbacher H, Bizu V, Nickola M, Wewetzer G, Wewetzer C, Ivarsson T, Skokauskas N, Wolters LH, Skarphedinsson G, Weidle B, de Haan E, Torp NC, Compton SN, Calvo R, Lera-Miguel S, Haigis A, Renner TJ, Conzelmann A. Internet-based cognitive behavioral therapy in children and adolescents with obsessive compulsive disorder: a feasibility study. J Neural Transm (Vienna). 2021 Sep;128(9):1445-1459. doi: 10.1007/s00702-021-02409-w. Epub 2021 Aug 25. PMID 34432173
- [Derived] Klein CS, Seyboth L, Conzelmann A, Schroder PA, Alt AK, Pascher A, Renner TJ, Gawrilow C, Hollmann K. Moderators of Symptom Self-Ratings in Pediatric Patients with Obsessive-Compulsive Disorder During a Digital Sensor-Assisted Treatment. Child Psychiatry Hum Dev. 2025 Nov 14. doi: 10.1007/s10578-025-01924-1. Online ahead of print. PMID 41236692
- [Derived] Alt AK, Klein CS, Pascher A, Conzelmann A, Kosel F, Kuhnhausen J, Hollmann K, Renner TJ. Acceptance of a sensor-based online psychotherapy for adolescents with obsessive-compulsive disorder (SSTeP-KiZ). Digit Health. 2025 Mar 28;11:20552076251327046. doi: 10.1177/20552076251327046. eCollection 2025 Jan-Dec. PMID 40162174
- [Derived] Klein CS, Alt AK, Pascher A, Kuhnhausen J, Seizer L, Ilg W, Thierfelder A, Primbs J, Menth M, Barth GM, Gawrilow C, Conzelmann A, Renner TJ, Hollmann K. Cognitive behavioral therapy for pediatric obsessive-compulsive disorder delivered via internet videoconferencing: a manualized sensor-assisted feasibility approach. Child Adolesc Psychiatry Ment Health. 2024 Dec 4;18(1):154. doi: 10.1186/s13034-024-00844-7. PMID 39633405
- [Derived] Klein CS, Hollmann K, Kuhnhausen J, Alt AK, Pascher A, Seizer L, Primbs J, Ilg W, Thierfelder A, Severitt B, Passon H, Worz U, Lautenbacher H, Bethge WA, Lochner J, Holderried M, Swoboda W, Kasneci E, Giese MA, Ernst C, Barth GM, Conzelmann A, Menth M, Gawrilow C, Renner TJ. Lessons learned from a multimodal sensor-based eHealth approach for treating pediatric obsessive-compulsive disorder. Front Digit Health. 2024 Sep 24;6:1384540. doi: 10.3389/fdgth.2024.1384540. eCollection 2024. PMID 39381777